CLINICAL TRIAL: NCT01117779
Title: Tracking Renal Tumors After Cryoablation Evaluation (TRACE) Registry
Brief Title: Tracking Renal Tumors After Cryoablation Evaluation
Acronym: TRACE
Status: Terminated | Type: Observational
Why Stopped: Boston Scientific acquisition of BTG/Galil Medical - business decision made to stop follow-up early
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CUC10-RNL02
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Kidney Neoplasms
Keywords: kidney tumors; renal tumors; renal cell carcinoma; kidney lesions; renal lesions; cryoablation; cryotherapy; cryosurgery
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Kidney lesions amenable to cryoablation: Kidney lesions treated with cryoablation.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  Other Names: Visual-ICE cryoablation system; SeedNet cryoablation system; PresIce cryoablation system; IceRod cryoablation needle; IceRod PLUS cryoablation needle; IceRod CX cryoablation needle; IceEDGE 2.4 cryoablation needle; IceSphere cryoablation needle

SUMMARY:
TRACE is an observational, open-label, single-arm, multi-center registry of subjects who have undergone renal lesion cryoablation per their physician's standard of care. Patients 18 years of age or older who have been determined to be an appropriate candidate for cryoablation will be offered enrollment into the registry. Subjects will be observed for five years from the date of their cryoablation procedure.

DETAILED DESCRIPTION:
The registry is non-interventional; it will neither direct the cryoablation procedures performed nor define the post-surgery follow-up of each subject. A subject's participation in the registry will not influence or direct subject treatment procedures or follow-up care. Physicians will use their discretion and personal standards of care to select subjects, perform the cryoablation procedures and define appropriate follow-up visit schedules for their subjects; it is anticipated that subjects will be seen at least once per year during the five-year follow-up period of TRACE. Subjects may be followed by the physician performing the cryoablation procedure or by their local/personal physician. The enrolling physician will be responsible for providing the follow-up data to the registry and will, as appropriate, work with a subject's local/personal physician to collect the follow-up data.

ELIGIBILITY:
Suggested Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has a renal lesion suspicious for malignancy.
* Patient is to undergo renal lesion cryoablation via a Galil Medical cryoablation system using Galil Medical needles for treatment of primary or recurrent disease.
* Patient is to be available for long-term follow-up per the enrolling physician's standard care practices.
* Patient has provided written informed consent.

Suggested Exclusion Criteria:

* Patient is either currently using or has used within the last 30 days an investigational product of any type.
* Patient has metastatic disease to or from the kidney.
* Patient has had previous therapy on the index lesion (e.g. radiofrequency, cryoablation, partial nephrectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Academic medical centers and community-based physicians
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Savage, MD, Study Chair — Medical University of South Carolina; Peter Clark, MD, Study Chair — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - University of California Irvine, Orange, California
  - Kaiser Permanente, Denver, Colorado
  - University of Kentucky, Lexington, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldfarb HA. Nd:YAG laser laparoscopic coagulation of symptomatic myomas. J Reprod Med. 1992 Jul;37(7):636-8. PMID 1387912
- [Background] Saliken JC, Donnelly BJ, Rewcastle JC. The evolution and state of modern technology for prostate cryosurgery. Urology. 2002 Aug;60(2 Suppl 1):26-33. doi: 10.1016/s0090-4295(02)01681-3. PMID 12206845
- [Background] Rewcastle JC, Sandison GA, Saliken JC, Donnelly BJ, McKinnon JG. Considerations during clinical operation of two commercially available cryomachines. J Surg Oncol. 1999 Jun;71(2):106-11. doi: 10.1002/(sici)1096-9098(199906)71:23.0.co;2-z. PMID 10389867
- [Background] Rewcastle JC, Hahn LJ, Saliken JC, McKinnon JG. Use of a moratorium to achieve consistent liquid nitrogen cryoprobe performance. J Surg Oncol. 1997 Oct;66(2):110-3. doi: 10.1002/(sici)1096-9098(199710)66:23.0.co;2-g. PMID 9354166
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Finley DS, Beck S, Box G, Chu W, Deane L, Vajgrt DJ, McDougall EM, Clayman RV. Percutaneous and laparoscopic cryoablation of small renal masses. J Urol. 2008 Aug;180(2):492-8; discussion 498. doi: 10.1016/j.juro.2008.04.019. Epub 2008 Jun 11. PMID 18550087

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryoablation: Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  There were a total of 246 ITT participants out of that 145 participants had lesion biopsy with proven Renal Cell Carcinoma (RCC).
Period: Overall Study
Arm/Group | Cryoablation
Started | 246
Completed | 246
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cryoablation: Participants with kidney lesions treated with cryoablation.
  Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  There were a total of 246 ITT participants with 145 of those having lesion(s) with biopsy proven Renal Cell Carcinoma (RCC).
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 240
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 203
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 246
Lesion Size [Median (Inter-Quartile Range); unit: cm] — Lesion size measured by greatest trans-axial diameter (cm)
  cm | 2.5 [2.0 to 3.1]
Quality of Life (QOL) Over time as assessed by the Short Form-12 (SF-12) GM [Median (Full Range); unit: score on a scale] — QoL SF12 is a health status survey to monitor outcomes in general and specific populations. Scoring system for the SF12 is norm based scoring (NBS).This rescaling is done by linear transformation.The scale for each component is provided where the min = worst health and max= best health. Scale range (min-max,range) : GH 23.9-63.7,39.8; PF 25.6-57.1,31.5 ; RP 23.6-57.5, 33.9 ; BP 21.7-57.7,36.1 ; VT 29.4-68.7, 39.4 ; SF 21.3-56.9,35.6; RE 14.7-56.3,41.6; HM 18.3-64.2,45.9;PCS 9.9-76,66 MCS 3.2-77.9,74.7
  score on a scale
    General Health | 47.750 [33.84 to 57.69]
    Physical Functioning | 49.190 [41.32 to 57.06]
    Role Physical | 49.000 [40.54 to 57.46]
    Bodily Pain | 48.710 [39.69 to 57.73]
    Vitality | 49.070 [39.23 to 58.90]
    Social Functioning | 48.010 [39.11 to 56.90]
    Mental Health | 52.740 [41.26 to 58.47]
    Role Emotional | 56.280 [40.69 to 56.28]
    Physical Component Summary | 46.930 [38.23 to 54.64]
    Mental Component Summary | 52.72 [44.11 to 57.53]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Lesion Size
Description: Changes to lesion size using greatest trans-axial diameter (cm) from baseline through the follow-up intervals.
Time Frame: Baseline and months 6, 12, 24, 36, 48 and 60
Population: Participants for whom cryoablation via GALIL Medical Cryoablation system was performed with available data at the respective time point.
Measure: Median (Inter-Quartile Range); unit: cm
Units Other Than Participants: lesions
Groups:
- Cryoablation: Patient with kidney lesions treated with cryoablation.
  Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance.
  There were a total of 246 ITT patients with 145 patients had biopsy proven Renal Cell Carcinoma (RCC).
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
Number analyzed (lesions) | 252
cm
  Baseline | 2.5 [2.0 to 3.1]
  Month 6 | -0.2 [-0.7 to 0.4]
  Month 12 | -0.4 [-0.9 to -0.1]
  Month 24 | -0.8 [-1.6 to -0.2]
  Month 36 | -1.0 [-1.8 to -0.5]
  Month 48 | -1.0 [-1.7 to -0.4]
  Month 60 | -1.0 [-1.8 to -0.4]

2. Primary Outcome: Renal Function Status
Description: Determined by the estimated Median Glomerular Filtration Rate (eGFR) measure using mL/min
Time Frame: Baseline and months 6, 12, 24, 36, 48 and 60
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
ml/min
  Baseline | 64.9 [50.6 to 81.8]
  Month 6 | 60.3 [48.3 to 78.3]
  Month 12 | 59.75 [47.5 to 73.7]
  Month 24 | 59.72 [42.3 to 75.3]
  Month 36 | 57.51 [43.3 to 73.4]
  Month 48 | 59.50 [47.0 to 70.5]
  Month 60 | 60.00 [43.9 to 74.5]

3. Primary Outcome: Hospital Stay
Description: Length of time in hospital is the duration of the patient's in-hospital time measured in hours, from intervention to discharge with the average duration of hospitalization being 2 days but could be much longer.
Time Frame: Average duration of 2 days or longer
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
hours | 29.3 [25.8 to 34.1]

4. Primary Outcome: Post-cryoablation Lesion Recurrence With Enhancement
Description: Lesions with imaging that showed contrast enhancement based on investigator assessment.
Time Frame: Months 6, 12, 24, 36, 48 and 60
Population: Lesion recurrence with enhancement
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
Number analyzed (lesions) | 248
lesions
  Month 6 | 4
  Month 12 | 3
  Month 24 | 4
  Month 36 | 1
  Month 48 | 4
  Month 60 | 1

5. Primary Outcome: Disease-specific Survival Rates
Description: Disease-specific survival rate is the time in days from cryoprocedure to death due to kidney cancer. Subjects who are alive will be censored at date of their last visit. Subjects who have died from causes other than kidney cancer will be censored at the time of death. Patients are followed up for duration of registry which is 5 years.
Time Frame: Month 60
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
Participants
  Alive | 221
  Death due to other causes | 25

6. Primary Outcome: Overall Survival Rates
Description: Death due to any cause
Time Frame: Month 60
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
Participants
  Not censored (death) | 25
  Censored | 221

7. Primary Outcome: Quality of Life Assessment
Description: QoL SF12 is a health status survey to monitor outcomes in general and specific populations. Scoring system for the SF12 is norm-based scoring (NBS). This rescaling is done by linear transformation.The scale for each component is provided where the min = worst health and max= best health. Scale range (min-max,range): GH 23.9-63.7,39.8; PF 25.6-57.1,31.5 ; RP 23.6-57.5, 33.9; BP 21.7-57.7,36.1; VT 29.4-68.7, 39.4; SF 21.3-56.9,35.6; RE 14.7-56.3,41.6; HM 18.3-64.2,45.9; PCS 9.9-76,66 MCS 3.2-77.9,74.7
Time Frame: Months 6 and 12
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 234
score on a scale
  General Health at month 6 | 47.750 [33.84 to 57.69]
  General Health at month 12 | 47.750 [33.84 to 57.69]
  Physical Functioning at month 6 | 41.320 [33.45 to 57.06]
  Physical Functioning at month 12 | 49.190 [41.32 to 57.06]
  Role Physical at month 6 | 44.770 [40.54 to 57.46]
  Role Physical at month 12 | 49.000 [40.54 to 57.46]
  Bodily Pain at month 6 | 48.710 [39.69 to 57.73]
  Bodily Pain at month 12 | 48.710 [39.69 to 57.73]
  Vitality at month 6 | 49.070 [39.23 to 58.90]
  Vitality at month 12 | 49.070 [39.23 to 58.90]
  Social Functioning at month 6 | 48.010 [39.11 to 56.90]
  Social Functioning at month 12 | 48.010 [39.11 to 56.90]
  Mental Health at month 6 | 52.740 [41.26 to 58.47]
  Mental Health at month 12 | 52.740 [41.26 to 58.47]
  Role Emotional at month 6 | 51.080 [40.69 to 56.28]
  Role Emotional at month 12 | 51.080 [35.49 to 56.28]
  Physical Component Summary at month 6 | 44.990 [35.49 to 54.26]
  Physical Component Summary at month 12 | 45.690 [37.69 to 56.64]
  Mental Component summary at month 6 | 52.720 [44.11 to 57.53]
  Mental Component summary at month 12 | 52.320 [43.64 to 57.38]

8. Primary Outcome: Development of Metastatic Disease.
Description: Time between cryotherapy and first evidence of metastatic disease
Time Frame: Month 60
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
months | 18.7 [10 to 44.8]

9. Primary Outcome: Total Number of Recurrences
Description: Total recurrences based on imaging with enhancement and retreatments (eg: nephrectomy, partial nephrectomy or ablation).
Time Frame: Month 60
Measure: Number; unit: recurrence
Arm/Group | Cryoablation
Number analyzed (Participants) | 246
recurrence | 18

10. Secondary Outcome: Procedure Method Outcomes
Description: An assessment of outcomes across laparoscopic-assisted, percutaneous and open cryoablation procedures.
Time Frame: During the procedure and immediately after it, an average of 2 hours.
Population: Participants treated with laparoscopic, percutaneous, or open procedure.
Measure: Number; unit: participants
Groups:
- INTENT TO TREAT (ITT)- POPULATION; RENAL CELL CARCINOMA (RCC) POPULATION: Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  There were a total of 246 ITT participants with 145 of those having lesion(s) with biopsy proven Renal Cell Carcinoma (RCC).
Arm/Group | INTENT TO TREAT (ITT)- POPULATION | RENAL CELL CARCINOMA (RCC) POPULATION
Number analyzed (Participants) | 246 | 145
participants
  Procedure Method: Laparoscopic | 99 | 63
  Procedure Method: Percutaneous | 146 | 81
  Procedure Method: Open | 1 | 1
  Number of lesions treated with cryoablation is One | 242 | 144
  Number of lesions treated with cryoablation is Two | 2 | 1
  Number of lesions treated with cryoablation is Three | 2 | 0
  Type of hemostatic agents or maneuvers used is None | 154 | 85
  Type of hemostatic agents or maneuvers used=Compression | 6 | 3
  Type of hemostatic agents or maneuvers used=Suturing | 4 | 2
  Type of hemostatic agents or maneuvers used=Floseal | 74 | 48
  Type of hemostatic agens or maneuvers used=Surgical | 79 | 52
  Type of hemostatic agents or maneuversed used=Other | 2 | 2
  Method of monitoring iceball formation=CT | 145 | 80
  Method of monitoring iceball formation=Ultrasound | 100 | 64
  Number of freeze/thaw cycles=0* | 1 | 1
  Number of freeze/thaw cycles=2 | 228 | 133
  Number of freeze/thaw cycles=3 | 12 | 9
  Number of freeze/thaw cycles=4 | 5 | 2
  Complications (malfunction of cryoablation system) | 3 | 3
  Intra-operative patient complications | 13 | 9

11. Secondary Outcome: Standard of Care Follow-up Procedures
Description: Characterization of standards of care for cryoablation procedure follow-up across the participating registry centers.
Time Frame: These outcomes are measured at each follow-up visit out to 5 years post-cryo procedure
Population: Is participant disease free (renal specific?) Are there new therapies for renal cancer (patient specific)
Measure: Number; unit: participants
Groups:
- ITT Population; RCC Population: Participants with kidney lesions treated with cryoablation.
  Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  There were a total of 246 ITT participants with 145 of those having lesion(s) with biopsy proven Renal Cell Carcinoma (RCC).
Arm/Group | ITT Population | RCC Population
Number analyzed (Participants) | 246 | 145
participants
  Disease free=Yes | 114 | 61
  Disease free=No | 8 | 7
  Disease free=Indeterminate | 2 | 2
  New therapies for renal cancer (patient specific)=Yes | 4 | 4
  New therapies for renal cancer (patient specific)=Yes [Local] | 4 | 4
  New therapies for renal cancer (patient specific)=Yes [Systemic] | 0 | 0
  New thereapies for renal cancer (patient specific)=No | 121 | 67

ADVERSE EVENTS:
Time Frame: Median follow-up of 60.1 months
Description: Potentially and directly related cryoablation AEs, SAEs/UADEs
Groups:
- Kidney Lesions Amenable to Cryoablation [ITT Population]: Kidney lesions treated with cryoablation.
  Cryoablation: Cryoablation (freezing) with Galil Medical cryoablation systems and needles under imaging guidance
  There were a total of 246 ITT patients with 145 patients having lesions biopsied and proven Renal Cell Carcinoma (RCC).
Arm/Group | Kidney Lesions Amenable to Cryoablation [ITT Population]
All-Cause Mortality (participants affected / at risk) | 26/246
Serious Adverse Events (participants affected / at risk) | 11/246
Other Adverse Events (participants affected / at risk) | 33/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kidney Lesions Amenable to Cryoablation [ITT Population] (N=246)
BLEEDING/HEMORRHAGE, GU (Surgical and medical procedures) | 2 (2)
ARRHYTHMIA-SUPRAVENTRICULAR (Cardiac disorders) | 1 (1)
HEMATOMA (Surgical and medical procedures) | 1 (1)
INFECTION (DOCUMENTED CLINICALLY) WITH GRADE 3 OR 4 ANC (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL HEMORRHAGE (Renal and urinary disorders) | 1 (1)
STRICTURE OF THE COLLECTION SYSTEM OR URETERS/STRICTURE/STENOSIS (Renal and urinary disorders) | 1 (1)
OTHER (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kidney Lesions Amenable to Cryoablation [ITT Population] (N=246)
OTHER (General disorders) | 10 (10)
PAIN (General disorders) | 7 (7)
HEMATOMA (Surgical and medical procedures) | 6 (6)
CREATININE ELEVATION (Renal and urinary disorders) | 4 (4)
URINARY RETENTION/OLIGURIA (Renal and urinary disorders) | 4 (4)
BLEEDING/HEMORRHAGE, GU (Renal and urinary disorders) | 2 (2)
VOMITING (General disorders) | 2 (2)
ARRHYTHMIA-SUPRAVENTRICULAR (Cardiac disorders) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BLEEDING/HEMORRHAGE, GI (Gastrointestinal disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL HEMORRHAGE (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the Boston Scientific (BSCI) Clinical Trial Agreement, BSCI needs to publish first.

PIs may publish their own data one year after the study has completed. If the PI wishes to publish after BSCI, then BSCI needs to be acknowledged in the publication.

DOCUMENTS (2):
  • Study Protocol (2011-05-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT01117779/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT01117779/SAP_001.pdf